CLINICAL TRIAL: NCT06593899
Title: The Total Neoadjuvant Therapy for Hypofractionated Radiotherapy Combined with AI Regimens in Soft Tissue Sarcoma of the Extremities: a Phase 2 Single Arm Multicenter Study
Brief Title: The Total Neoadjuvant Therapy for Soft Tissue Sarcoma of the Extremities
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Yong Yang, DR., Fujian Medical University Union Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRGHO-STS23
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-12

CONDITIONS: Soft Tissue Sarcomas
MeSH Terms: conditions — Sarcoma | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypofractionated Radiotherapy (Experimental): The patients in the study underwent a 1-week course of hypofractionated radiotherapy. Following the completion of radiotherapy, chemotherapy with the AI regimen (doxorubicin + ifosfamide) was initiated one week later. The AI regimen chemotherapy was administered for a duration of 9 weeks. Subsequently, surgery was scheduled to commence 1-2 weeks after the completion of chemotherapy.
  Interventions: Radiation: Hypofractionated Radiotherapy; Drug: 3 cycles of AI

INTERVENTIONS:
Radiation: Hypofractionated Radiotherapy — Hypofractionated radiotherapy Preoperative hypofractionated 5x5 Gy radiotherapy (5 consecutive days) prescribed on planned target volume
Drug: 3 cycles of AI — Three courses of doxorubicin and ifosfamide (AI, doxorubicin 75 mg/sqm and ifosfamide 10 g/sqm with prophylactic mesna)

SUMMARY:
For localized soft tissue sarcomas (STS) of the extremities, limb-sparing or conservative surgery with perioperative radiotherapy (RT) is the standard of care. However, several challenges persist. Notably, there are exceedingly high rates of distant metastatic recurrence even after surgical resection and RT, and conventional fractionated radiotherapy has a prolonged duration (5-6 weeks). With advancements in RT technology, the gradual expansion of hypofractionated radiotherapy regimens enables significantly shorter treatment durations. Promising recent reports on 1-week hypofractionated RT regimens, such as the 5X5 Gy RT regimens, have demonstrated reasonable local control and acceptable toxicity in resectable STS.Addressing the challenge of distant metastasis, previous studies have indicated that AI regimens are expected to eliminate micrometastases and improve survival in patients with STS at a high risk of distant relapse. Therefore, the goal of this clinical trial is to investigate whether hypofractionated RT combined with a sequential chemotherapy（AI regimens）can enhance short-term treatment efficacy for extremity STS patients without compromising local control rates and increasing related toxicities

ELIGIBILITY:
Inclusion Criteria:

1. Primary soft tissue sarcoma of the extremities, with one of the following characteristics: high grade, ≥5cm or deep tumor, the need for neoadjuvant radiotherapy was determined after multidisciplinary consultation.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2.
3. Age 18-75 years old.
4. Histologic diagnosis of soft tissue sarcoma.
5. Can tolerate radiotherapy and AI regimen treatment.
6. The function of major organs is normal.

Exclusion Criteria:

1. There were no patients with gross tumors after unplanned mass resection in another hospital.
2. Patients with other comorbidities cannot use AI chemotherapy: drug allergy, active bleeding, ulcers, intestinal perforation, intestinal obstruction, uncontrollable hypertension, grade III-IV cardiac insufficiency (NYHA standards), severe liver and renal insufficiency ( Level IV) etc.
3. New malignant tumors within 5 years (except cervical carcinoma in situ or early cutaneous basal cell carcinoma).
4. Pathological types: nonpleomorphic rhabdomyosarcoma, Ewing sarcoma.
5. Soft tissue sarcoma curable by simple expansion.
6. Previous history of radiotherapy to the same site.
7. Combined with distant metastasis (M1) or lymph node metastasis (N1).
8. Have other severe medical comorbidities that preclude surgery or participation in the study.
9. Previous exposure to chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of EORTC-STBSG classifications A-C (less than 10% tumour residual) | Surgery

SECONDARY OUTCOMES:
Postoperative wound complications | 3 months
Overall survival | 24 months after treatment completion
Local control | 24 months after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Yong Yang, Doctor, Principal Investigator — Director of the radiotherapy department
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blay JY, Honore C, Stoeckle E, Meeus P, Jafari M, Gouin F, Anract P, Ferron G, Rochwerger A, Ropars M, Carrere S, Marchal F, Sirveaux F, Di Marco A, Le Nail LR, Guiramand J, Vaz G, Machiavello JC, Marco O, Causeret S, Gimbergues P, Fiorenza F, Chaigneau L, Guillemin F, Guilloit JM, Dujardin F, Spano JP, Ruzic JC, Michot A, Soibinet P, Bompas E, Chevreau C, Duffaud F, Rios M, Perrin C, Firmin N, Bertucci F, Le Pechoux C, Le Loarer F, Collard O, Karanian-Philippe M, Brahmi M, Dufresne A, Dupre A, Ducimetiere F, Giraud A, Perol D, Toulmonde M, Ray-Coquard I, Italiano A, Le Cesne A, Penel N, Bonvalot S; NETSARC/REPPS/RESOS and French Sarcoma Group-Groupe d'Etude des Tumeurs Osseuses (GSF-GETO) Networks. Surgery in reference centers improves survival of sarcoma patients: a nationwide study. Ann Oncol. 2019 Jul 1;30(7):1143-1153. doi: 10.1093/annonc/mdz124. Erratum In: Ann Oncol. 2019 Aug 1;30(8):1407. doi: 10.1093/annonc/mdz170. PMID 31081028
- [Background] Gronchi A, Stacchiotti S, Verderio P, Ferrari S, Martin Broto J, Lopez-Pousa A, Llombart-Bosch A, Dei Tos AP, Collini P, Jurado JC, De Paoli A, Donati DM, Poveda A, Quagliuolo V, Comandone A, Grignani G, Morosi C, Messina A, De Sanctis R, Bottelli S, Palassini E, Casali PG, Picci P. Short, full-dose adjuvant chemotherapy (CT) in high-risk adult soft tissue sarcomas (STS): long-term follow-up of a randomized clinical trial from the Italian Sarcoma Group and the Spanish Sarcoma Group. Ann Oncol. 2016 Dec;27(12):2283-2288. doi: 10.1093/annonc/mdw430. Epub 2016 Oct 11. PMID 27733375
- [Background] Kalbasi A, Kamrava M, Chu FI, Telesca D, Van Dams R, Yang Y, Ruan D, Nelson SD, Dry SM, Hernandez J, Chmielowski B, Singh AS, Bukata SV, Bernthal NM, Steinberg ML, Weidhaas JB, Eilber FC. A Phase II Trial of 5-Day Neoadjuvant Radiotherapy for Patients with High-Risk Primary Soft Tissue Sarcoma. Clin Cancer Res. 2020 Apr 15;26(8):1829-1836. doi: 10.1158/1078-0432.CCR-19-3524. Epub 2020 Feb 13. PMID 32054730
- [Background] Gobo Silva ML, Lopes de Mello CA, Aguiar Junior S, D'Almeida Costa F, Stevanato Filho PR, Santoro Bezerra T, Nakagawa SA, Nascimento AG, Werneck da Cunha I, Spencer Sobreira Batista RM, Nicolau Daher UR, Da Cruz Formiga MN, Germano JN, Catin Kupper BE, De Assis Pellizzon AC, Lopes A. Neoadjuvant hypofractionated radiotherapy and chemotherapy for extremity soft tissue sarcomas: Safety, feasibility, and early oncologic outcomes of a phase 2 trial. Radiother Oncol. 2021 Jun;159:161-167. doi: 10.1016/j.radonc.2021.03.033. Epub 2021 Mar 31. PMID 33798613